CLINICAL TRIAL: NCT07272369
Title: Comparison of the Effect of Video-Assisted Teaching and Web-Based Game on Teaching Intramuscular Injection to Nursing Students
Brief Title: Video vs. Game-Based Teaching of Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nehir Demirel, Öğr. Gör. Dr., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NehirAlev
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Gamification; Video-Based Learning; Students, Nursing; Intramuscular Injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Based Teaching (Experimental)
  Interventions: Other: Video Based Teaching of Intramuscular Injection
- Game-Based Teaching (Experimental)
  Interventions: Other: Game-Based Teaching of Intramuscular Injection

INTERVENTIONS:
Other: Video Based Teaching of Intramuscular Injection — Video Based Teaching of Intramuscular Injection
  Arms: Video Based Teaching
Other: Game-Based Teaching of Intramuscular Injection — Game-Based Teaching of Intramuscular Injection
  Arms: Game-Based Teaching

SUMMARY:
One of the psychomotor skills that must be taught to nursing students is intramuscular injection (IME), which is frequently used among parenteral drug administration techniques and is associated with a higher incidence of medical errors. Incorrect injection techniques can lead to serious complications such as nerve damage, tissue trauma, and infection. It is critically important for nursing students to learn this skill correctly in order to ensure patient safety and improve their clinical skills. Therefore, it is essential to use different teaching methods in nursing education, especially in acquiring and developing IME skills. Games, a common type of virtual simulation, are pedagogical tools that offer students extensive learning opportunities and enjoyable teaching through the use of interactive media. Video-supported teaching is also a powerful tool for acquiring clinical skill proficiency. However, no research has been found comparing the effectiveness of web-based games and video-supported teaching in determining the effectiveness of intramuscular training. Furthermore, students' test anxiety is an important factor that should not be overlooked and that hinders learning. Therefore, this project proposal is planned as a fully experimental design with the aim of comparing the effects of two different teaching methods on intramuscular injection application skill levels and test anxiety levels in the teaching of intramuscular injection application. In this context, the Student Introduction Form, IME Skill Checklist, and Revised Test Anxiety Scale will be used to collect data.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Being a first-year nursing student
* Taking the Fundamentals of Nursing course for the first time
* Having no communication problems related to vision or hearing
* Volunteering to participate in the study

Exclusion Criteria:

* Being a graduate of a Health Vocational High School
* Being a transfer student who has previously received training on intramuscular injection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Intramuscular Injection Skill Performance Score | 2 month
  Skill performance will be evaluated using the Intramuscular Injection Skill Checklist (0-100 points)

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No